CLINICAL TRIAL: NCT06152523
Title: Monalizumab and MEDI5752 in Patients With MSI and/or dMMR Metastatic Cancer
Acronym: MONAMI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP220097; 2022-004122-22 (EudraCT Number)
Record Dates: First submitted 2023-09-05; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: MSI; dMMR Colorectal Cancer
Keywords: Cancer; MSI/dMMR tumors; Monalizumab; MEDI5257; Efficacy; Safety/tolerability; Pharmacokinetic; MSI phenotype; Immune Checkpoint Inhibitors; Immunotherapy; Cytotoxic chemotherapy
MeSH Terms: conditions — Neoplasms | interventions — monalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSI/dMMR tumors across all solid tumor types in adult patients (Experimental)
  Interventions: Drug: Monalizumab/MEDI5257

INTERVENTIONS:
Drug: Monalizumab/MEDI5257 — Phase II trial using an A'Hern design with a safety lead-in cohort to assess the safety/tolerability of the combination of monalizumab and MEDI5752 in patients with metastatic MSI/dMMR cancer

SUMMARY:
MSI is a molecular indicator of defective DNA mismatch repair (dMMR). The MSI/dMMR status is observed in all tumor types, representing notably 5% of metastatic colorectal cancers (mCRC), 25% of advanced endometrial cancer and 8% of metastatic gastric cancer.

MSI/dMMR cancers are highly immunogenic. MSI/dMMR tumors are characterized by a high tumor mutational burden with highly immunogenic neoantigens. These tumors are associated with an upregulation of immune checkpoints (PD1, PDL1, CTLA4, etc.) that protects MSI cancer cells from their hostile immune micro-environment, characterized by a high infiltration of activated cytotoxic T CD8+ and NK lymphocytes. Consequently, MSI/dMMR cancers are highly sensitive to ICIs, whatever the tumor location. MSI/dMMR status is a predictive biomarker for the efficacy of immunotherapy, regardless of the tumor type. Then, by several phase II and III studies The efficacy of immunotherapy has been demonstrated as front-line treatment for patients with chemotherapy-naive MSI/dMMR mCRC and gastric cancer. The phase III KEYNOTE-177 trial evaluating first-line treatment of pembrolizumab in patients with MSI/dMMR mCRC demonstrated its superiority over first-line chemotherapy, with a significant improvement of health-related quality of life. At final analysis, the median follow-up was 44.5 months. Median PFS was 16.5 versus 8.2 months (HR = 0.59; 95%CI 0.45-0.79). The hazard ratio favored pembrolizumab versus chemotherapy with a trend toward reduction in the risk of death (HR 0.74; 95% CI, 0.53-1.03; P=0.0359), despite a 60% effective crossover rate. Pembrolizumab has been approved by the FDA and the EMA for patients with newly diagnosed MSI/dMMR mCRC and is now the standard of care for this population. Also, the phase III CHECKMATE-649 trial reveal that the Combination of immunotherapy and cytotoxic chemotherapy is the new standard of care for patients with newly diagnosed metastatic oesogastric cancer. Importantly, results of the CHECKMATE-649 are outstanding for the subgroup population of MSI/dMMR gastric cancer patients (N = 44). Indeed, the unstratified hazard ratio for OS with nivolumab plus chemotherapy versus chemotherapy alone was 0.33 (95% CI 0.12-0.87) for patients with MSI/dMMR tumors. All in all, ICIs are the standard of care in first-line setting for patients with mCRC or metastatic oesogastric cancer. Besides, several phase II studies suggest that ICI combinations might overcome primary resistance to anti-PD1 monotherapy These data justify the development of bispecific monoclonal antibodies targeting both PD1 and CTLA4 such as MEDI5752. MEDI5752 has been developed based on the observation that there is a higher expression of PD-1/CTLA-4 on tumor resident versus peripheral T cells. Preclinical data show MEDI5752 fully suppresses PD-1 and preferentially inhibits CTLA-4 in the tumor versus the periphery, which is meant to uncouple CTLA-4 dependant peripheral toxicity from antitumor activity Natural killer cells are integral to the functioning of the innate immune system and play an important role in innate antitumor immunity. There is a growing body of evidence for targeting the NKG2A/HLA-E axis in combination with other ICIs to sensitize tumors to ICI therapy. NKG2A recognizes the non-classical HLA class I molecule HLA-E. The NKG2A receptor is found on peripheral NK cells and subsets of T cells in cancer patients. It is also present in tumor-infiltrating NK and cytotoxic T cells. Importantly, NK cells and the NKG2A/HLA-E axis play a crucial role in MSI/dMMR tumors. Therefore, a combined blockade of non-redundant checkpoint pathways to unleash NK and T cells seems particularly promising for MSI/dMMR neoplasms. Monalizumab specifically binds and blocks the inhibitory receptor NKG2A. Monalizumab has been investigated in combination with ibrutinib (in chronic lymphoid leukemia), cetuximab +/- durvalumab (in squamous cell carcinoma of the head and neck, and in solid tumors), durvalumab +/- FOLFOX (in solid tumors). In the first-in-human dose escalation of monalizumab plus durvalumab, a manageable toxicity profile was shown.

Taken together, these data provide a strong rational to combine an inhibitor of the NKG2A/HLA-E axis with a bispecific monoclonal antibody targeting both PD1 and CTLA4 for patients with metastatic MSI/dMMR cancers.

DETAILED DESCRIPTION:
MONAMI is a multicenter (4 French hospitals) single-arm phase II trial according to A'Hern's design with a safety lead-in. For the achievement of the main objectif and primary endpoint, the tumor measurements using CT-scan (preferred option) or MRI will be performed at baseline, 6 weeks, 12 weeks, 18 weeks and 24 weeks. The same type of imaging (CT or MRI) as the one used at baseline will have to be performed for all tumor imaging evaluation.

The study contains a safety lead-in (N = 9) in which the safety and tolerability of monalizumab plus MEDI5752 will be assessed after the second cycle (the first 42 days of treatment).

The Data Safety Monitoring Board (DSMB) will evaluate the safety data at pre-specified intervals (every 4 weeks and at the end of the safety lead-in) and at additional points during the conduct of the safety lead-in, if necessary. The tolerability assessment will be based upon occurrence of dose-limiting toxicities. Additional patients will be enrolled based on assessments of the safety data by the DSMB during the safety lead-in Enrollment will be put on hold after the inclusion of the first patient in the safety lead-in until the end of the DLT period and until a discussion with the DSMB can occur. After every 3 new included patients in the safety lead-in until the end of the DLT period of the last included patient and until a discussion with the DSMB can occur. During this period, if 3 patients experience dose-limiting toxicities until a discussion with the DSMB can occur and after the inclusion of all the patients of the safety lead-in, until the end of the DLT period of the last patient and until a discussion with the DSMB can occur for the authorization to initiate the second part of the phase II study.

Patients will be treated with monalizumab 750 mg and MEDI5752 750 mg every 3 weeks intravenously, for 32 infusions (or less in case of RECIST disease progression or limiting toxicity, whichever occurs first).

Monalizumab will be supplied by AstraZeneca as a lyophilized product for concentrate for solution for infusion MEDI5752 will be supplied by AstraZeneca as a lyophilized product for concentrate for solution for infusion

Because of the possibility of an initial increase in tumor burden caused by immune-cell infiltration in the setting of a T-cell response (termed "pseudoprogression") with cancer immunotherapy, radiographic progression per RECIST v1.1 may not be indicative of true disease progression. During the study, participants who meet criteria for disease progression per RECIST v1.1 (unconfirmed disease progression per iRECIST criteria: iuPD) and show evidence of clinical benefit may continue study treatment at the Investigator's discretion provided that the participants meet all of the following criteria:

* Absence of clinically important symptoms and signs (including worsening of laboratory values) indicative of disease progression
* Investigator-assessed potential clinical benefit for the participant
* The participant is tolerating study drugs
* No decline in ECOG Performance Status
* Absence of rapid progression of disease or of progressive tumor at critical anatomical sites (e.g., cord compression) requiring urgent alternative medical intervention For participants receiving treatment beyond progression, an additional radiographic assessment/scan should be performed within 6 weeks of initial progression to determine whether there has been a stabilization or decrease in the tumor size or continued PD (confirmed disease progression per iRECIST criteria; icPD). Study treatment should be discontinued permanently upon documentation of further progression.

Safety lead-in cohort : 9 Phase II study : 29 Total : 43 patients maximum

* 38 evaluable patients
* If necessary, inclusions may be continued to reach the required number of evaluable patients within the limit of 5 additional participants

Duration of enrolment period (including safety lead-in cohort with interruption of inclusion after the first 9 participants): 2 years

The length of participation for participants, of which:

* Maximum period between screening and treatment initiation: 21 days
* Treatment duration: 2 years maximum
* Duration of follow-up period: 3 years from inclusion in the study Total study duration: 5 years and 21 days

Patients included in the safety lead-in will be analyzed as part of the overall population of the phase II study

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria :

1. Signed and dated patient informed consent form (ICF) and willingness to comply with all study procedures and availability for the study duration,
2. Age ≥ 18 years,
3. Body weight > 35 kg,
4. Eastern Cooperative Oncology Group performance status of 0 or 1,
5. Life expectancy ≥ 12 weeks,
6. Histologically confirmed carcinoma,
7. dMMR and/or MSI tumor status defined by:

   * Loss of MMR protein expression using immunohistochemistry with four (anti-MLH1, anti-MSH2, anti-MSH6, and anti-PMS2) antibodies,
   * and/or ≥ two instable markers by polymerase chain reaction using standard panels; if two instable markers in the pentaplex panel, it is required to present confirmation of the dMMR status by immunohistochemistry or a comparison of the tumor PCR test with matched to normal tissue.
8. Documented advanced or metastatic disease not suitable for complete surgical resection,
9. Prior treatment for metastatic disease: patients are eligible if they have progressed on or following prior treatment and who have no satisfactory alternative treatment options , except for patients :

   * with MSI/dMMR colorectal or oesogastric cancer who are eligible for study enrollment even if they did not receive prior treatment for metastatic disease,
   * with advanced or recurrent endometrial carcinoma, who are eligible for study enrollment if they have disease progression on or following prior treatment with a platinum-containing therapy in any setting and who are not candidates for curative surgery or radiation
   * with unresectable or metastatic small intestine or biliary cancer, who are eligible for the study enrolment if they have disease progression on or following at least one prior therapy
10. At least one measurable lesion as assessed by CT-scan or magnetic resonance imaging (MRI) according to RECIST v1.1 and feasibility of repeated radiological assessments. Participants with lesions in a previously irradiated field as the sole site of measurable disease will be permitted to enroll provided the lesion(s) have demonstrated clear progression and can be measured accurately,
11. Availability of a representative tumor specimen for exploratory translational research; tumor tissue specimens, either formalin-fixed, paraffin-embedded (FFPE) tissue block or unstained tumor tissue sections (minimum of 30 positively charged slides) from primary or metastatic site must be submitted to the central laboratory,
12. Baseline-corrected QT interval < 470 ms
13. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:

    * Hematological status:

      * White blood cell > 2000/µL;
      * Neutrophils > 1500/µL;
      * Platelets > 100.000/µL;
      * Hemoglobin > 9.0 g/dL;
    * Adequate renal function:

    Serum creatinine level < 150 µM and calculated creatinine clearance (Cockcroft-Gault) ≥ 45 mL/minute,

    - Adequate liver function:
    * Serum bilirubin ≤ 1.5 x upper normal limit (ULN) or direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN;
    * Alkaline phosphatase (ALP) ≤ 3 x ULN;
    * Alanine aminotransferase (ALT) ≤ 3.0 x ULN;
    * Aspartame aminotransferase (AST) ≤ 3.0 x ULN;
    * Prothrombin time (PT)/International normalized ratio (INR) and partial PT (PTT) ≤ 1.5 x ULN unless participants are receiving anticoagulant therapy and their INR is stable and within the recommended range for the desired level of anticoagulation,
14. Females of childbearing potential:

    - Must have negative pregnancy test at screening , prior to each administration of investigational product and at each follow-up visit until 140 days after last treatment;
    * If sexually active with a nonsterilized male partner, must use at least one highly effective method of birth control from screening to 140 days after the last dose of MEDI5752 and monalizumab;
    * IT IS STRONGLY RECOMMENDED THAT nonsterilized male partners of female subjects of childbearing potential use a male condom plus spermicide from screening to 140 days after the last dose of MEDI5752 (Note: Male condoms are not reliable as a sole contraception method)
    * Refer to APPENDIX 18.1 : Definition of Women of Childbearing Potential for definitions of females of childbearing potential
15. Female subjects must not breastfeed and must not donate, or retrieve for their own use, ova from screening to 140 days after the last dose of MEDI5752 and monalizumab
16. Nonsterilized male subjects who are sexually active with a female partner of childbearing potential must use a condom with spermicide from screening to 140 days after the last dose of MEDI5752 and monalizumab (Note: Male condoms are not reliable as a sole contraception method). IT IS STRONGLY RECOMMENDED THAT female partners of a male subject also use at least one highly effective method of contraception throughout this period. In addition, male subjects must refrain from fathering a child or donating sperm during the study and for 140 days after the last dose of MEDI5752 and monalizumab.
17. Registration in a national health care system (AME are not allowed).

Exclusion Criteria:

Exclusion Criteria :

1. Active brain metastases or known leptomeningeal metastases.
2. Persistence of toxicities related to prior chemotherapies grade > 1 (NCI CTCAE v5.0; except alopecia, fatigue, or peripheral sensory neuropathy, which can be grade 2),
3. Concomitant unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, radiotherapy, immunotherapy),
4. Major surgical procedure within 4 weeks prior to initiation of study treatment,
5. More than 3 prior lines of chemotherapy,
6. Prior treatment with an anti-PD1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways, including prior therapy with anti-tumor vaccines or other immuno-stimulatory antitumor agents,
7. Patients receiving any investigational drug within the previous 21 days before study treatment,
8. Impossibility of submitting to the medical follow-up of the study for geographical, social or psychic reasons,
9. Patients with an active, known or suspected autoimmune disease. Can be enrolled: Patients with type I diabetes mellitus, hypothyroidism requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger,
10. History of interstitial lung disease or pneumonitis,
11. Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to treatment initiation.

    Treatment permitted in the absence of active autoimmune disease: Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent.,
12. Prior malignancy active within the previous 3 years except for except for:

    * Locally curable cancers that have been apparently cured (e.g. squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast),
    * Lynch syndrome-related cancer in complete remission for > 1 year;
13. Evidence of the following infections:

    * Active infection including tuberculosis (TB) (clinical evaluation that includes clinical history, physical examination, and radiographic findings and TB testing in line with local practice),
    * or human immunodeficiency virus (HIV) (positive for HIV-1 or HIV-2 antibodies),
    * or active or uncontrolled hepatitis B (HBV) or hepatitis C (HCV). Participants are eligible if they:

      * Have controlled hepatitis C viral load defined as undetectable hepatitis C RNA by PCR either spontaneously or in response to a successful prior course of anti-hepatitis C therapy,
      * Have received HBV vaccination with only anti-HBs positivity and no clinical signs of hepatitis,
      * Are HBsAg- and anti-HBc+ (ie, those who have cleared HBV after infection) and meet conditions i-iii below:
      * Are HBsAg+ with chronic HBV infection (lasting 6 months or longer) and meet conditions i-iii below:

    HBV DNA viral load <100 IU/mL Have normal transaminase values, or, if liver metastases are present, abnormal transaminases, with a result of AST/ALT <3 × ULN, which are not attributable to HBV infection Start or maintain antiviral treatment if clinically indicated as per the investigator.

    - or active hepatitis A (refer to Section 5.7 for screening tests)
14. Prior allogeneic bone marrow transplantation or prior solid organ transplantation,
15. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, cardiomyopathy of any etiology, symptomatic congestive heart failure (as defined by New York Heart Association class > 2), uncontrolled hypertension, unstable angina pectoris, history of myocardial infarction within the past 12 months, cardiac arrhythmia, ILD, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the subject to give written informed consent,
16. Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of the subject's safety or study results
17. Known allergy/hypersensitivity to any component or excipients of study agents,
18. Administration of a (attenuated) live vaccine within 30 days of planned start of study therapy of known need for this vaccine during treatment,
19. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 140 days after the last dose of Monalizumab and MEDI5752
20. Patient on tutelage or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities | Day 42 / 3 years
Assess the objective response rate (ORR) per RECIST v.1.1 criteria at 24 weeks of monalizumab and MEDI5752 in combination in patients with MSI/dMMR metastatic cancer (Phase II study) | Week 24

SECONDARY OUTCOMES:
Incidence and severity of adverse events graded according to the NCI CTCAE version 5.0 | 3 Years
Incidence and severity of adverse events of special interest graded according to the NCI CTCAE version 5.0, version | 3 Years
Incidence of dose interruptions, dose modifications and discontinuations due to adverse events | 3 Years
Objective response rate per RECIST v.1.1 criteria at 24 weeks since the initiation of the treatment, defined by the number of patients with partial or complete response at 24 weeks (Phase II Study) | Week 24
Assess the safety profile of MEDI5752 plus monalizumab (adverse events per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.5.0) ( (Phase II Study) | Week 24
Assess ORR per RECIST v.1.1 at 48 and 96 weeks and iRECIST at 24, 48 and 96 weeks with MEDI5752 and monalizumab (Phase II Study) | Week 24, Week 48, Week 96
Assess progression-free survival per RECIST v.1.1 and iRECIST at 24, 48 and 96 weeks with MEDI5752 and monalizumab (Phase II Study) | Week 24, Week 48, Week 96
Assess overall survival at 24, 48 and 96 weeks with MEDI5752 and monalizumab (Phase II Study) | Week 24, Week 48, Week 96
Concentration max (Cmax) of monalizumab | Week 3, Week 6, Week 18, Week 30, Week 54, Week 96
Concentration min (Cmin) of monalizumab | Week 3, Week 6, Week 18, Week 30, Week 54, Week 96
Concentration max (Cmax) of MEDI5752 | Week 3, Week 6, Week 18, Week 30, Week 54, Week 96
Concentration min (Cmin) of MEDI5752 | Week 3, Week 6, Week 18, Week 30, Week 54, Week 96
Concentration (Cmin) of MEDI5752 | Week 3, Week 6, Week 18, Week 30, Week 54, Week 96
Frequency of antidrug antibody development | Week 3, Week 6, Week 18, Week 30, Week 54, Week 96
Rate of misdiagnosed MSI/dMMR tumors as centrally evaluated by immunohistochemistry and/or molecular methods (Phase II Study) | Week 6, Week 9, Week 27
Tumor response as evaluated by RECIST and iRECIST criteria (Phase II Study) | Week 2, Week 6, Week 12, Week 18, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96, Week 108, Week 120, Week 132, Week 144, Week 156
Progression free survival assessed by RECIST and iRECIST criteria (Phase II Study) | Week 2, Week 6, Week 12, Week 18, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96, Week 108, Week 120, Week 132, Week 144, Week 156
Overall survival (OS) (Phase II Study) | Week 148
  OS is defined as the time between beginning of treatment and death from any cause. Survival data will be censored at the last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Romain COHEN, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Department of medical oncology - Saint-Antoine Hospital, Paris, France